CLINICAL TRIAL: NCT07332429
Title: Evaluation of the Efficacy and Safety of Alcovit (Zeolite Clinoptilolite) in Reducing Blood Alcohol Concentration in Healthy Individuals
Brief Title: Efficacy and Safety of Alcovit in Reducing Blood Alcohol Concentration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galzu Institute of Research, Teaching, Science and Applied Technology (Other)
Collaborators: Hospital Santa Casa de Misericordia de Campos (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IGZ-06
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Drinking; Blood Alcohol Content; Hangover
Keywords: Zeolite Clinoptilolite; Alcovit; Alcohol Absorption; Medical Device; Hangover Prevention; Blood Alcohol Concentration
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Four parallel groups with 1:1:1:1 randomization comparing Alcovit® (zeolite clinoptilolite) versus placebo, administered at different time points relative to alcohol consumption. Group 1: Alcovit® administered 2-3 minutes before standardized alcohol intake. Group 2: Alcovit® administered within 5 minutes after completing alcohol intake. Group 3: Placebo administered 2-3 minutes before alcohol intake. Group 4: Placebo administered within 5 minutes after completing alcohol intake. Each participant remains in their assigned group throughout the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alcovit (Pre-consumption) (Experimental): Participants receive the investigational device immediately before (2-3 minutes) consuming the standardized alcohol dose.
  Interventions: Device: Alcovit® (Zeolite Clinoptilolite)
- Alcovit (Post-consumption) (Experimental): Participants receive the investigational device immediately after (maximum 5 minutes) consuming the standardized alcohol dose.
  Interventions: Device: Alcovit® (Zeolite Clinoptilolite)
- Placebo (Pre-consumption) (Placebo Comparator): Participants receive the placebo immediately before consuming the standardized alcohol dose.
  Interventions: Device: Placebo
- Placebo (Post-consumption) (Placebo Comparator): Participants receive the placebo immediately after consuming the standardized alcohol dose.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Alcovit® (Zeolite Clinoptilolite) — Effervescent powder for oral suspension presented in 15g sachets, containing zeolite clinoptilolite (approximately 96% of the formulation) associated with B-complex vitamins (B1, B6, B12), vitamin C, and cupric chlorophyllin as natural colorant. The device is administered either immediately before alcohol consumption (2-3 minutes prior) or immediately after alcohol consumption (maximum 5 minutes after) depending on the assigned study arm.
  Other Names: Alcovit (Pre-consumption); Alcovit (Post-consumption)
  Arms: Alcovit (Post-consumption); Alcovit (Pre-consumption)
Device: Placebo — Effervescent powder for oral suspension presented in 15g sachets. Inert substance with identical appearance, taste, and texture to Alcovit®, but without the active ingredient (zeolite clinoptilolite). The placebo is administered either immediately before alcohol consumption (2-3 minutes prior) or immediately after alcohol consumption (maximum 5 minutes after) depending on the assigned study arm.
  Other Names: Placebo (Pre-consumption); Placebo (Post-consumption)
  Arms: Placebo (Post-consumption); Placebo (Pre-consumption)

SUMMARY:
The goal of this clinical trial is to learn if Alcovit® (zeolite clinoptilolite) works to reduce blood alcohol concentration in healthy adults aged 18-70 years who are occasional or moderate alcohol consumers. It will also learn about the safety and tolerability of Alcovit®. The main questions it aims to answer are:

* Does Alcovit® reduce blood alcohol concentration when administered before or after standardized alcoholic beverage consumption compared to placebo?
* What is the rate of alcohol elimination from the blood (mg/dL/hour) in participants taking Alcovit® compared to placebo?
* Is Alcovit® well tolerated when administered before or after alcohol consumption?

Researchers will compare Alcovit® administered before alcohol consumption, Alcovit® administered after alcohol consumption, placebo administered before alcohol consumption, and placebo administered after alcohol consumption to see if Alcovit® effectively reduces blood alcohol levels.

Participants will:

* Consume a standardized alcoholic beverage under controlled conditions;
* Take Alcovit® or a placebo either 2-3 minutes before or after (within 5 minutes) alcohol consumption;
* Have blood samples collected at baseline (30 minutes before), and at 20, 40, and 60 minutes after alcohol consumption to measure blood alcohol concentration;
* Complete breathalyzer (etilometer) measurements at the same time points;
* Answer questionnaire to assess alcohol hangover severity;
* Have safety blood tests performed to monitor liver and kidney function.

DETAILED DESCRIPTION:
The product has extensive international experience, having been marketed in several countries (Germany, Poland, Romania, Russia, Australia, Mexico, Colombia, Croatia, United States, Ukraine and Sweden) over the past 15 years, totaling 1,387,500 sachets sold without reports of toxicity.

The safety of clinoptilolite zeolite has been extensively evaluated by the European Food Safety Authority (EFSA) and by clinical trials, which confirmed its safety at typical food exposure levels, with no toxic side effects observed in humans or animals, even with prolonged use.

Alcovit® is formulated as an effervescent powder for suspension presented in 15g sachets and intended for healthy adults who are occasional or moderate consumers of alcoholic beverages.

The mechanism of action of Alcovit® is based on the ability of clinoptilolite zeolite to adsorb alcohol molecules in the stomach and small intestine, preventing their systemic absorption and promoting their natural elimination through the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 70 years;
* Occasional or moderate alcohol consumers;
* Willing to abstain from alcohol and Alcovit® for a period established in the study;
* Voluntary willingness to participate in the study and sign the Informed Consent Form (ICF);
* Availability to comply with the study schedule.

Exclusion Criteria:

* History of alcohol use disorder (alcoholism) or abuse of other illicit substances;
* Hepatic, renal, gastrointestinal diseases, diabetes, and chronic conditions;
* Use of medications that interact with alcohol, including but not limited to: non-steroidal anti-inflammatory drugs (NSAIDs such as ibuprofen, diclofenac, naproxen), analgesics, antibiotics, antidepressants, benzodiazepines, anticoagulants, or any other medication that may interfere with alcohol metabolism or increase risks associated with alcohol consumption;
* Pregnancy or breastfeeding (beta-hCG test will be performed);
* Known allergy to any component of Alcovit® or placebo;
* Patients already enrolled in other clinical trials;
* Inability to provide free and informed consent;
* Any clinically significant medical condition or medical history that, in the investigator's opinion, may discourage participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2026-05-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Blood Alcohol Levels and Breathalyzer Readings - Pre-consumption Administration | Baseline (30 minutes before), 20 minutes, 40 minutes, and 60 minutes after alcohol consumption (Day 1)
  Analysis of the reduction in blood alcohol levels and breathalyzer (ethylometer) readings in the Alcovit® group compared to the placebo group before alcohol consumption.
Reduction in Blood Alcohol Levels and Breathalyzer Readings - Post-consumption Administration | Baseline (30 minutes before), 20 minutes, 40 minutes, and 60 minutes after alcohol consumption (Day 1).
  Analysis of the reduction in blood alcohol levels and breathalyzer (ethylometer) readings in the Alcovit® group compared to the placebo group after alcohol consumption.

SECONDARY OUTCOMES:
Correlation Between Blood Alcohol Reduction and Breathalyzer Readings | Baseline (30 minutes before), 20 minutes, 40 minutes, and 60 minutes after alcohol consumption (Day 1)
  Correlation between the reduction in blood alcohol levels and breathalyzer (ethylometer) readings.
Correlation Between Elimination Rate in Blood and Breathalyzer | Baseline (30 minutes before), 20 minutes, 40 minutes, and 60 minutes after alcohol consumption (Day 1).
  Correlation between the elimination rate of alcohol in blood and breathalyzer (ethylometer) readings.
Hangover Symptom Severity Using AHSS | 24 hours after alcohol consumption (Day 1)
  Evaluation of Alcovit® efficacy in mitigating hangover symptoms using the total score and subdomains of the Alcohol Hangover Severity Scale (AHSS).
Participant Experience with Alcovit® (Patient-Reported Outcomes) | Day 1 to Day 2
  Participant experience with Alcovit® assessed by participant questionnaire.
Adverse Events Reported by Participants (Clinician-Reported Outcomes) | Baseline (30 minutes before), 20 minutes, 40 minutes, and 60 minutes after alcohol consumption (Day 1)
  Analysis of adverse events reported by participants.
Number and Type of Adverse Events (Clinician-Reported Outcomes) | Day 1 to Day 44 (6 weeks)
  Number and type of adverse events, unexpected adverse events, and serious adverse events.
Changes in Hepatic Function Markers (Clinician-Reported Outcomes) | Day 1 to Day 44 (6 weeks)
  Changes in hepatic function between Alcovit® administration groups before and after alcohol ingestion (distilled and fermented beverages) compared to control for AST, ALT, GGT, alkaline phosphatase (ALP), total bilirubin and fractions.
Changes in Renal Function Markers (Clinician-Reported Outcomes) | Day 1 to Day 44 (6 weeks)
  Changes in renal function between Alcovit® administration groups before and after alcohol ingestion (distilled and fermented beverages) compared to control for urea, creatinine, electrolytes, and urinalysis.
Ease of Handling and Administration (Clinician-Reported Outcomes/Patient-Reported Outcomes) | Day 1.
  Ease of handling and administration of Alcovit® assessed by questionnaire administered to nursing staff.
Baseline Population Characteristics (Clinician-Reported Outcomes) | Day 1 (baseline)
  Characterization of the study population and identification of potential confounding factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santa Casa de Misericórdia de Campos, Campos dos Goytacazes, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality in accordance with Brazilian data protection laws (LGPD - Lei Geral de Proteção de Dados) and ethical requirements. Study results will be published in aggregated form only.